CLINICAL TRIAL: NCT06949527
Title: Ultrasonographic and Sonoelastographic Evaluation of the Effects of Open Bite Activator and Anterior Skeletal Anchorage-Supported Vertical Elastics on the Masseter Muscle in Skeletal Open Bite Cases
Brief Title: Effects of Open Bite Activator and Skeletal Anchorage-Supported Vertical Elastics on the Masseter Muscle
Acronym: OB-MUSCLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murat Kaan Erdem (Other)
Responsible Party: Sponsor-Investigator, Murat Kaan Erdem, PhD, DDS, Ankara University
Organization: Ankara University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANK-DHF-OBM-2025; 36290600/78 (Other: Ankara University Faculty of Dentistry Clinical Research Ethics Committee)
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Hyperdivergent Facial Pattern; Skeletal Open Bite; Hyperdivergent Growth Pattern; Anterior Open Bite
Keywords: Open Bite Treatment; Masseter Muscle; Ultrasound Imaging; Sonoelastography; Skeletal Anchorage; Vertical Elastics; Functional Orthodontic Appliance; Cephalometric Analysis
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Intervention Model Description: Participants received treatment with an open bite activator combined with vertical elastics supported by anterior skeletal anchorage in a single group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Functional Appliance with Skeletal Anchorage-Supported Vertical Elastics (Experimental): Patients were treated using a custom-made open bite activator combined with vertical elastics supported by anterior miniscrews placed between lateral and canine teeth in both jaws. The elastics applied 150g of force bilaterally and were worn for 20-22 hours per day over a 12-month period. The goal was to manage vertical skeletal development and evaluate changes in masseter muscle morphology via ultrasound and sonoelastography.
  Interventions: Device: Open Bite Activator with Skeletal Anchorage-Supported Vertical Elastics

INTERVENTIONS:
Device: Open Bite Activator with Skeletal Anchorage-Supported Vertical Elastics — A custom-made acrylic open bite activator was fabricated for each participant, with the bite registered 3-4 mm above freeway space. Miniscrews were placed between the lateral and canine teeth in both jaws. Vertical elastics (150g force) were applied bilaterally between miniscrews and the appliance. The intervention aimed to reduce vertical growth in posterior regions and stimulate anterior dentoalveolar development while improving masseter muscle morphology.
  Other Names: Functional Appliance; Vertical Elastics; Mini-Implants

SUMMARY:
This clinical trial aims to evaluate the effects of a combined treatment involving an open bite activator and anterior skeletal anchorage-supported vertical elastics on the masseter muscle in children with skeletal open bite. A total of 24 growing individuals with increased vertical skeletal pattern were treated with a functional appliance and intermaxillary vertical elastics supported by miniscrews placed in the anterior region. Ultrasonographic and sonoelastographic assessments were performed at baseline, 6 months, and 12 months to measure changes in masseter muscle thickness and stiffness. Cephalometric radiographs were also used to evaluate dentofacial structural changes. This study aims to provide insight into the soft tissue changes associated with functional orthopedic treatment in hyperdivergent patients.

DETAILED DESCRIPTION:
This prospective clinical study investigates the dentofacial and muscular effects of a combined orthopedic treatment method in patients with skeletal open bite. The intervention includes the use of an open bite activator appliance along with anterior skeletal anchorage-supported vertical elastics. The study was conducted at Ankara University Faculty of Dentistry, Orthodontics Department, and received ethical approval (Approval No: 36290600/78).

A total of 24 growing individuals (14 females, 10 males) with increased vertical facial pattern (GoGn/SN ≥ 36°) were treated over a 12-month period. Patients received custom-made open bite activators designed to eliminate occlusal contact in the anterior region and redirect functional forces posteriorly. Miniscrews were placed between the lateral and canine teeth in both the maxilla and mandible, and vertical elastics were applied between these skeletal anchorage points with a force of 150 grams on each side, worn for 20-22 hours daily.

Masseter muscle changes were assessed using ultrasonography and sonoelastography at three time points: baseline (T0), interim (6 months, T1), and end of treatment (12 months, T2). Muscle thickness and stiffness (elasticity) were measured bilaterally during rest and maximal clenching. Cephalometric radiographs were obtained at T0 and T2 to evaluate skeletal and dentoalveolar changes, including SNA, SNB, ANB angles, overbite, U1-PP, L1-MP, and other relevant vertical and angular measurements.

Statistical analysis revealed significant increases in masseter muscle thickness during the treatment period, especially between T0 and T1. Stiffness values peaked at T1 and slightly decreased at T2, but remained higher than baseline. Cephalometric findings showed improvements in overbite and reductions in vertical growth tendencies, including significant changes in GoGn/SN and PP-MP angles.

This study demonstrates that combined functional appliance and skeletal anchorage-based vertical control therapy can positively influence muscle structure and dentofacial morphology in hyperdivergent skeletal open bite cases. Ultrasonography and sonoelastography proved to be reliable, non-invasive methods for assessing soft tissue changes in orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

* GoGn/SN angle ≥ 36°
* Decreased overbite (dental open bite)
* In active growth phase (confirmed by hand-wrist radiograph)
* Good oral hygiene
* No prior orthodontic or orthognathic treatment

Exclusion Criteria:

* Presence of systemic disease or craniofacial deformity
* Poor oral hygiene
* Non-compliance with appliance wear
* Previous use of skeletal anchorage devices

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Change in masseter muscle thickness measured by ultrasonography | Baseline, 6 months, and 12 months
  Masseter muscle thickness (in millimeters) will be measured at rest and during maximal clenching using ultrasonography at three time points: baseline (T0), 6 months (T1), and 12 months (T2).

SECONDARY OUTCOMES:
Change in masseter muscle stiffness assessed by sonoelastography | Baseline, 6 months, and 12 months
  The ratio of stiff (red) areas to total cross-sectional area of the masseter muscle will be evaluated using shear wave sonoelastography at T0, T1, and T2.

CONTACTS AND LOCATIONS:
Overall Officials: Murat K Erdem, PhD, DDS, Principal Investigator — Ankara University
Locations (1):
- Ankara University Faculty of Dentistry, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data (IPD) may be shared upon reasonable request. No personal or identifiable information will be included in the shared data.